CLINICAL TRIAL: NCT02932852
Title: Autologous Adipose-Derived Adult Stem Cell Transplantation for Corneal Diseases
Acronym: A-ADAS-CT-CD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Collaborators: Reviva Pharmaceuticals (Industry); Hospital Universitario La Paz (Other); LASER VISION CENTER IN LIBANON (Unknown); OPTICA GENERAL IN LIBANON (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTP-007/15
Record Dates: First submitted 2016-10-02; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Hereditary Corneal Dystrophy; Keratoconus
Keywords: stem cell; mesenchymal; ADASc; transplantation; cornea; corneal defects; keratoconus; scaffold; lamina
MeSH Terms: conditions — Corneal Dystrophies, Hereditary; Keratoconus; Corneal Diseases | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GROUP I (Active Comparator): lipoaspiration and transplantation of ADAS alone without scaffold
  Interventions: Procedure: Lipoaspiration; Procedure: Transplantation
- GROUP II (Active Comparator): Lipoaspiration and transplantation of scaffold (human corneal decellularized lamina) without ADAS
  Interventions: Procedure: Lipoaspiration; Procedure: Transplantation
- GROUP III (Active Comparator): Lipoaspiration and transplantation of ADAS cellularized on scaffold (the human corneal decellularized lamina)
  Interventions: Procedure: Lipoaspiration; Procedure: Transplantation

INTERVENTIONS:
Procedure: Lipoaspiration — The patient will have a liposuction surgery from which the autologous ADAS cell to transplant in the cornea will be obtained.
Procedure: Transplantation — The ophthalmologist will carry out the transplantation of the ADAS cells with or without scaffold in the intrastromal cornea of the patient

SUMMARY:
Transplantation of cellularized human cornea impregnated and populated by mesenchymal stem cells derived from the patient's adipose tissue. The purpose of the study is to assess the safety, tolerability, and preliminary efficacy of transplantation of a single dose of autologous mesenchymal adipose tissue derived adult stem cells (ADAS) cellularized into laminas for subjects with corneal defects. 3 groups will be included in the study: (1) transplantation of ADAS alone without scaffold, (2) transplantation of scaffold (human corneal decellularized lamina) without ADAS, and (3) transplantation of ADAS cellularized on scaffold (the human corneal decellularized lamina)

DETAILED DESCRIPTION:
Different types of stem cells have been used in various ways in several research projects in order to find the optimal procedure to regenerate the human corneal stroma. It included several approaches which can be classified as intrastromal implantation of stem cells (1) alone, (2) together with a biodegradable scaffold, (3) with a non-biodegradable scaffold, or (4) with a decellularized corneal stromal scaffold. In fact, the complex structure of the corneal stroma has not been yet replicated, and there are well known drawbacks to the use of synthetic scaffold-based designs. Recently, several corneal decellularization techniques have been described, which provide an acellular corneal extracellular matrix (ECM). These scaffolds have gained attention in the last few years as they provide a more natural environment for the growth and differentiation of cells when compared with synthetic scaffolds. In addition, components of the ECM are generally conserved among species and are tolerated well even by xenogeneic recipients. Keratocytes are essential for remodeling the corneal stroma and for normal epithelial physiology. This highlights the importance of transplanting a cellular substitute together with the structural support (acellular ECM) to undertake these critical functions in corneal homeostasis. To the best of the investigators knowledge, all attempts to repopulate decellularized corneal scaffolds have used corneal cells, but these cells have major drawbacks that preclude their autologous use in clinical practice (damage of the donor tissue, lack of cells and inefficient cell subcultures), thus the efforts to find an extraocular source of autologous cells. A recent study by the investigators has shown a perfect biointegration of human decellularized corneal stromal sheets (100µm thickness) with and without h-ADASC colonization inside the rabbit cornea in vivo, without observing any rejection response despite the graft being xenogeneic. The investigators also demonstrated the differentiation of h-ADASCs into functional keratocytes inside these implants in vivo, which then achieved their proper biofunctionalization. According to the investigator's opinion the transplant of stem cells together with decellularized corneal ECM would be the best technique to effectively restore the thickness of a diseased human cornea, like in keratoconus. Through this technique, and using extraocular mesenchymal stem cells from patients, it is possible to transform allergenic grafts into functional autologous grafts, theoretically avoiding the risk of rejection.

The process flow is defined as following: (1) the file study: which start by receiving the file of the patient, the file will be forwarded to appointed physicians coordinators for review and submission of medical report, then the medical report will be evaluated within the cell therapy committee and the patient will be asked for clinical examination, and after consultation a reply to the patient with medical decision will follow with an approval or not to be recruited and if yes, a brief report about the procedure will be submitted and explained in details to the patient, a consent form must be signed if the patient agree to be included in the study, (2) the patient admission: which may start by completion of the procedure forms and doing the pre-op evaluation (initial work up defined as a clinical and biological assessment upon C.A.S which may include unaided and best spectacle corrected visual acuity, refraction, slit lamp examination, intraocular pressure, fundoscopy, corneal topography, aberrometry, endothelial cell count (specular microscopy) as well as blood tests) by an ophthalmologist, followed by lipoaspiration of the subcutaneous adipose tissue to be performed by a plastic surgeon, then sample processing at a cGMP facility for isolation and characterization of the stromal vascular fraction enriched with ADAS as well as laminas preparing (the quality control assessment will be realized before and after all the steps of the procedure starting from the ADAS collection to transplantation including cell culture, cell quiescence, decellularization of human corneal lamina, recellularization of the laminas with ADAS, and transplantation; the assessment will include cell viability, cell number, cell apoptosis, immunophenotyping, infection, inflammation by analyzing the secreted cytokines from ADAS, lamina cutting, lamina thickness, immunostaining, confocal microscopy, etc.); (3) the delivery (transplantation) which starts by a peribulbar or retrobulbar anesthesia where the patient is placed under operating microscope, followed by a femtosecond laser assisted mid-stromal lamellar dissection, then the ADAS or laminas or recellularized laminas will be placed within the pocket, and finally closed by a superior incision closure. The patient will be putted under antibiotic/steroids for a defined period and followed by the team at 1 week, 2 weeks, 1 month, 3 months, 6 months and 1 year.

This protocol of cell therapy will be applied exclusively at Laser Vision (Hazmieh-Lebanon) and prepared at Reviva Regenerative Medicine Center in affiliation with VISSUM (Alicante-Spain) and Optica General (Saida-Lebanon).

The patient's recruitment will take place: for the lipoaspiration, processing, preparing the celluraized laminas and quality control assessments, at the Middle East Institute of Health the Reviva Center (Bsalim-Lebanon) under the regulations of the hospital and the Reviva Center; for injection, at Laser vision (Hazmieh-Lebanon); and for follow-up, at Laser vision & optica general. All these steps are managed by VISSUM (Prof. J. ALIO).

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by corneal stromas dystrophies of any type, but particularly keratoconus, showing clear evidence at the ophthalmic examination of the presence and clear expression of the disease
* Age : ≥ 18 years
* Gender: any
* Willing to collaborate and to attend to the clinical follow ups for the next five years
* Patients willing to sign informed consent
* Able and willing to comply with all study requirements
* Patients with and no worse than 0.6 for the better vision patients
* Comprehensive clinical ophthalmological including slit lamp photography of the cornea of either eye
* Corneal topography map including both anterior and posterior corneal surfaces
* Specular microscopy
* Confocal microscopy of the centre of the cornea
* Absence of anterior segment inflammation
* Medically suitable to undergo corneal graft surgery with local anesthesia
* Medically suitable for general anesthesia or waking sedation, if needed
* Normal serum chemistry and hematology screening tests
* Negative human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV) serology
* No history of malignancy
* Complete history & physical examination
* Negative chest roentgenogram (CXR)
* Negative urinalysis (U/A)
* Normal thyroid exam

Exclusion Criteria:

* - Patients not willing to sign informed consent
* Defects in corneal transparency with a potential to affect the visual outcome
* Vision of 0.05 or less
* Severe corneal deformation
* Infection
* Moderate or severe dry eye
* Chronic ocular surface inflammation of any origin
* Previous ocular surgery other than cataract
* Presence of cataract or other media opacity that would influence ocular fundus documentation and adequate ERG and visual field evaluation.
* Other ophthalmic comorbidity like glaucoma and uveitis
* Known allergy: example to propacaine, ciprofloxacin, fluorescein , indocyanine green, or others to specify
* Known coagulation abnormalities
* Any medical condition likely interferes to cause serious adverse events during the study
* Presence of active or inactive choroidal neovascularization (CNV) in the eye to be treated
* History of malignancy
* History of cognitive impairments or dementia which may impact the patient's ability to participate in the informed consent process and to appropriately complete evaluations
* Any immunodeficiency
* Any current immunosuppressive therapy other than intermittent or low dose corticosteroids
* Renal insufficiency, as defined by creatine level >1.3 mg/dL.
* Serologic evidence of infection with Hepatitis B, Hepatitis C, or HIV
* If female, pregnancy or lactation.
* Any other medical condition, which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromises patient safety, or interferes with the interpretation of the study results.corneal dystrophies of any type, in a stage which either could be prevented in progression (with best corrected visual acuity superior to 0.6) or with indication for keratoplasty (best corrected visual acuity <0.2). The cases should not have defects in corneal transparency which would lead to vision of 0.05 or less or severe corneal optical deformation (in the case of keratoconus).
* The visual acuity of the eye to receive the transplant will be no better than 20/400
* The visual acuity of the eye in the better vision cohort to receive the transplant will be no better than 0.1 at the Snellen charts
* The visual acuity of the eye that is not to receive the transplant will be no better than 0.2 for the worse vision patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Vision recovery (Corrected Distance Visual Acuity) | post operative visit at 1 day, 1 month, 3 months and 6 months
  The Best Corrected Visual Acuity will be measured in each postoperative visit to control any important decrease relative to the surgery

SECONDARY OUTCOMES:
Corneal Thickness | post operative visit at 1 day, 1 month, 3 months and 6 months
  At each post operative visit a measurement of corneal pachymetry of the transplanted cornea will be carried out to detect any abnormal evolution
Topopgraphy | post operative visit at 1 month, 3 months and 6 months
  At each post operative visit a measurement of Anterior surface topography of the transplanted cornea will be carried out to detect any abnormal evolution
Anterior segment Optical Coherence Tomography | post operative visit at 1 month, 3 months and 6 months
  At each post operative visit a measurement anterior segment Optical Coherence Tomography of the transplanted cornea will be carried out to detect any abnormal evolution
Slit Lamp Observation | post operative visit at 1 day, 1 month, 3 months and 6 months
  At each post operative visit, the corneal aspect relative to new tissue will be evaluated by slit lamp observation
refraction measurement | post operative visit at 1 day, 1 month, 3 months and 6 months
  At each post operative visit, the corneal aspect relative to increase in irregular astigmatism will be evaluated by refraction measurement

CONTACTS AND LOCATIONS:
Overall Officials: Mona El Zarif, OD, Study Chair — Optica General
Locations (1):
- Optica General, Saida, Lebanon

REFERENCES:
- [Background] Alio del Barrio JL, Chiesa M, Garagorri N, Garcia-Urquia N, Fernandez-Delgado J, Bataille L, Rodriguez A, Arnalich-Montiel F, Zarnowski T, Alvarez de Toledo JP, Alio JL, De Miguel MP. Acellular human corneal matrix sheets seeded with human adipose-derived mesenchymal stem cells integrate functionally in an experimental animal model. Exp Eye Res. 2015 Mar;132:91-100. doi: 10.1016/j.exer.2015.01.020. Epub 2015 Jan 24. PMID 25625506
- [Background] De Miguel MP, Alio JL, Arnalich-Montiel F, Fuentes-Julian S, de Benito-Llopis L, Amparo F, Bataille L. Cornea and ocular surface treatment. Curr Stem Cell Res Ther. 2010 Jun;5(2):195-204. doi: 10.2174/157488810791268663. PMID 19941445
- [Background] Alio del Barrio JL, Chiesa M, Gallego Ferrer G, Garagorri N, Briz N, Fernandez-Delgado J, Sancho-Tello Valls M, Botella CC, Garcia-Tunon I, Bataille L, Rodriguez A, Arnalich-Montiel F, Gomez Ribelles JL, Antolinos-Turpin CM, Gomez-Tejedor JA, Alio JL, De Miguel MP. Biointegration of corneal macroporous membranes based on poly(ethyl acrylate) copolymers in an experimental animal model. J Biomed Mater Res A. 2015 Mar;103(3):1106-18. doi: 10.1002/jbm.a.35249. Epub 2014 Jun 18. PMID 24910285
- [Derived] Alio JL. Corneal regeneration: How can we make further progress in corneal surgery with advanced therapies to avoid corneal substitution: ESCRS Binkhorst Medal Lecture 2023. J Cataract Refract Surg. 2025 Nov 1;51(11):1026-1033. doi: 10.1097/j.jcrs.0000000000001745. PMID 41126474
- [Derived] El Zarif M, Alio JL, Alio Del Barrio JL, Abdul Jawad K, Palazon-Bru A, Abdul Jawad Z, De Miguel MP, Makdissy N. Corneal Stromal Regeneration Therapy for Advanced Keratoconus: Long-term Outcomes at 3 Years. Cornea. 2021 Jun 1;40(6):741-754. doi: 10.1097/ICO.0000000000002646. PMID 33591032